CLINICAL TRIAL: NCT04272437
Title: Concentrated Traditional Chinese Herbal Extract Granules TRA for Preventing Symptomatic Urinary Tract Infection Among High-risk Elderly Residing in Nursing Homes-A Randomized Placebo-Controlled Trial
Brief Title: TRA for Preventing Symptomatic Urinary Tract Infection Among High-risk Elderly Residing in Nursing Homes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Changhua Christian Hospital (Other)
Collaborators: Ministry of Health and Welfare, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MOHW107-CMAP-M-114-122113
Record Dates: First submitted 2020-02-10; First posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Urinary Tract Infections
Keywords: Nursing Homes; TCM herbal extracts
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to receive intervention or placebo.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants were randomly assigned to take either TRA or placebo. Participants in the two groups orally ingested one package of granules (5 g/package) two times daily after lunch and dinner. The placebo was prepared as granules by Chuang Song Zong Pharmaceutical Co., Ltd, and the packaging of the placebo was identical to that of herbal extract granules. During the trial, neither the care providers(including family numbers and nursing-home colleagues) nor investigators ( assist doctors or nurses ) were aware of the group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TRA group (Experimental): "Tokoro Combination" and "Rehmannia and Akebia Formula" (TRA) in each one batch number were manufactured by Chuang Song Zong Pharmaceutical Co., Ltd., a famous manufacturer of concentrated herbal extract granules in agreement with the standards of good manufacturing practices (GMP) in Kaohsiung City, Taiwan.
  TRA contains "Tokoro Combination" and "Rehmannia and Akebia Formula" "Tokoro Combination" and "Rehmannia and Akebia Formula" consists of Dioscorea Hypoglaucae Rhizoma, Acori Graminei Rhizoma, Linderae Radix, Alpiniae Oxyphyllae Fructus, Poria, Rehmanniae Radix, Akebiae Caulis, Lophatheri Hebra, and Glycyrrhizae Radix at a 2:2:2:2:1:1.3:1.3:1.3:2.5 ratio.
  Interventions: Drug: Concentrated herbal extract granules TRA
- placebo group (Placebo Comparator): The placebo was also prepared as granules by Chung Song Zong Pharmaceutical Co., Ltd., and the packaging of the placebo was identical to that of TRA.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Concentrated herbal extract granules TRA — Concentrated herbal extract granules Subjects in the TRA group orally ingested one package of granules (5 g/package) two times daily with warm water after lunch and dinner for 6 consecutive weeks.
  Arms: TRA group
Drug: Placebo — Subjects in the placebo group orally ingested one package of granules (5 g/package) two times daily with warm water after lunch and dinner for 6 consecutive weeks.
  Arms: placebo group

SUMMARY:
Urinary tract infection (UTI) is one of the most common infection in nursing home residents, and symptomatic UTI in the nursing home setting is the most frequent reason for hospitalization and antimicrobial therapy in Taiwan. Increasing antimicrobial resistance has stimulated interest in non-antibiotic prophylaxis of UTI. The primary aim of this study is to test the efficacy of standardized concentrated herbal extract granules TRA in the reduction of the incidence of symptomatic UTI and associated hospitalization in high-risk nursing home residents. These aims were accomplished by conducting a double-blind randomized placebo-controlled efficacy trial of TRA daily versus placebo granules in a cohort of Changhua County nursing home residents in Taiwan.

A total of 164 nursing home residents at high risk for UTI were be enrolled. A permuted block design with a block size of 6 were conducted. And a Stratification by nursing home accounted for potentially different standards of care. Subjects will be randomly assigned to receive either TRA (10 g) or the placebo two times per day for 42 consecutive days. All subjects in both groups will also continuously receive their daily medication without any dose or medicine change. Urinalysis was evaluated before and after administration. Independent statisticians performed the data analysis at the end of the trial.

DETAILED DESCRIPTION:
The standardized concentrated herbal extract granules TRA were the combination of "Tokoro Combination(Pi-Hsieh-Fen-Ching-Yin Extract Granules)" and "Rehmannia and Akebia Formula (Dao Chi San Extract Powder)". "Tokoro Combination" and "Rehmannia and Akebia Formula" in each one batch number were used, manufactured by Chuang Song Zong Pharmaceutical Co., Ltd., a famous GMP manufacturer of concentrated herbal extract granules in agreement with international standards. The TRA was prepared in small granules, including concentrated herbal extract granules of "Tokoro Combination"(50%) and "Rehmannia and Akebia Formula" (50%). Both medicines have already been approved by the Ministry of Health and Welfare in Taiwan as ethical drugs. TRA granules were packed in oblique glassine packages. The placebo was also prepared as granules by Chuang Song Zong Pharmaceutical Co., Ltd., and the packaging of the placebo was identical to that of TRA. The chemical composition of TRA was analyzed and profiled by using a high performance liquid chromatography (HPLC). The major components were diosgenin, yamogenin, betulin, oleanolic acid, hederagenin, akeboside, β-sitosterol, stigmasterol, inositol, catalpol, glycyrrhizin, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Nursing home residents;
2. 65 years or older; and
3. High UTI risk

   * Catheterization (>1 m/o),
   * Diabetes mellitus, or
   * At least one UTI in the preceding year.

Exclusion Criteria:

1. Not expected to be in the nursing home for at least one month (i.e. pending discharge, terminal life expectancy < 1 month);
2. On chronic suppressive antibiotic or anti-infective therapy
3. On dialysis for end stage renal disease; or
4. previous ADR to herbals.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 162 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-03-03 (Actual)

PRIMARY OUTCOMES:
Number of Episodes of Symptomatic UTI During Administration | 42 days
  Nursing home medical record and National Health Insurance(NHI) IC cards checking were both performed every week for the symptomatic UIT diagnosis and hospitalization recording. Suspected UTI episodes that were recorded in nursing home medical record were reviewed by chart review, symptoms, signs, and laboratory data were recorded, two investigators determined if the definition of symptomatic UTI was met.

SECONDARY OUTCOMES:
Number of Episodes of Symptomatic UTI Onset From First Administration Till 180 Days | 180 days.
  Nursing home medical record and National Health Insurance(NHI) IC cards checking were both performed every week for the symptomatic UIT diagnosis and hospitalization recording. Suspected UTI episodes that were recorded in nursing home medical record were reviewed by chart review, symptoms, signs, and laboratory data were recorded, two investigators determined if the definition of symptomatic UTI was met.
Accumulated Rate of Symptomatic UTI During Administration | 42 days.
  Nursing home medical record and National Health Insurance(NHI) IC cards checking were both performed every week for the symptomatic UIT diagnosis and hospitalization recording. Suspected UTI episodes that were recorded in nursing home medical record were reviewed by chart review, symptoms, signs, and laboratory data were recorded, two investigators determined if the definition of symptomatic UTI was met.
Accumulated Rate of Symptomatic UTI Onset From First Administration Till 180 Days | 180 days.
  Nursing home medical record and National Health Insurance(NHI) IC cards checking were both performed every week for the symptomatic UIT diagnosis and hospitalization recording. Suspected UTI episodes that were recorded in nursing home medical record were reviewed by chart review, symptoms, signs, and laboratory data were recorded, two investigators determined if the definition of symptomatic UTI was met.
The Change of Urinalysis From Baseline to 42 Days | 42 days
  Sterile urine specimen collection from a foley catheter or clean catch midstream urine for urinalysis were obtained from baseline to 6 weeks for each participant for study purposes.
  Changes in urine species were texted by using chemical strip and urine sediment method in the Department of Laboratory Medicine at ChungHua Christrian Hospital. The items for urinalysis were as following: specific gravity, pH value, protein, nitrite, WBC esterase, RBC( in high-power field), RBC( in high-power field), squamous epithelial cell( in high-power field), bacteria( in high-power field), etc.
Number of Deaths Onset From First Administration Till 180 Days | 180 days
  All-cause deaths were recorded.

OTHER OUTCOMES:
Number of Adverse Events in Participants | 42 days

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Traditional Chinese Medicine, Changhua Christian Hospital, Changhua, Taiwan